CLINICAL TRIAL: NCT05252624
Title: Impact of Henagliflozin on Cardiac Structure, Function and Biomarkers of Heart Failure in Patients With Persistent Atrial Fibrillation
Brief Title: Henagliflozin in Patients With Atrial Fibrillation
Acronym: HENA-AF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Chang sheng Ma, Director of Cardiology, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022-HENA
Record Dates: First submitted 2022-01-11; First posted 2022-02-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Atrial Fibrillation
Keywords: Heart Failure; SGLT2i; Cardiac structure; Cardiac function
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure | interventions — henagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: Henagliflozin (Active Comparator): Single 5 mg tablet, administered orally once daily for 6 months
  Interventions: Drug: Henagliflozin 5Mg Tab
- Placebo Comparator: Placebo (Placebo Comparator): Single 5 mg tablet, administered orally once daily for 6 months
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — Placebo tablet manufactured to mimic henagliflozin 5 mg tablet
  Arms: Placebo Comparator: Placebo
Drug: Henagliflozin 5Mg Tab — Single oral tablet
  Arms: Active Comparator: Henagliflozin

SUMMARY:
The HENA-AF trial will evaluate the effects of henagliflozin on cardiac structure, function, and biomarkers of HF in patients with AF. Participants with persistent AF, enlarged left atrium, and at least another cardiovascular risk factor will be randomized to henagliflozin or placebo. Cardiac MRI will be performed at baseline and at 6 months to measure the changes in cardiac structure and function. The primary hypothesis is that henagliflozin will reduce the left atrial volume index at 6 months in patients with AF.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is a major public health burden worldwide. Heart failure (HF) is one of the most common causes of death in patients with AF. Clinical trials have indicated that SGLT2i can reduce the risk of AF and HF in patients with diabetes, and improve the prognosis in patients with HF. However, whether SGLT2i can improve cardiac function and reduce the risk of HF in patients with AF remains unclear. The purpose of the HENA-AF trial is to evaluate the effects of henagliflozin on cardiac structure, function, and biomarkers of HF in patients with AF.

The HENA-AF trial will include approximately 100 persistent AF patients with enlarged left atrium and at least another cardiovascular risk factor. Participants will be randomized to henagliflozin or placebo. Cardiac MRI will be performed at baseline and at 6 months to measure the changes in cardiac structure and function. The primary hypothesis is that henagliflozin will reduce the left atrial volume index at 6 months in patients with AF.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 and ≤80 years old
2. Persistent AF: ECG or Holter diagnosed AF for more than 1 month
3. LA enlargement (LAAPD ≥40mm and <60mm)
4. One or more risk factors as follows: (1) ≥65 years old; (2) LVH: echocardiographic calculation of left ventricular mass index (LVMI) male ≥115g/m2; female ≥95g/m2 (LVMI=LVM/BSA,LVM=1.04 × [(LVID+IVST+LVPWT) 3-LVID3] * 0.8 * 0.6) BSA (m2) =0.0061 * height (cm) + 0.0128 * weight (kg)-0.1529; (3) Coronary heart disease (CHD): CHD diagnosed by coronary angiography or CTA, or previous history of myocardial infarction, or revascularization (PCI, CABG); (4) Peripheral artery disease (PAD): imaging examination (ultrasound, CTA, MRA or angiography) indicates carotid or lower extremity artery stenosis >50%. Or peripheral vascular revascularization (stent or endarterectomy); (5) Obesity: BMI ≥28

Exclusion Criteria:

1. Intention of catheter ablation of AF in the next 6 months
2. Cardiovascular events (myocardial infarction, etc.) or cardiac surgery in the past 3 months
3. Clinically diagnosed heart failure (objective evidence of elevated natriuretic peptide levels and/or cardiogenic pulmonary/systemic congestion on the basis of structural and/or functional abnormalities) or left ventricular ejection fraction (LVEF) <40%
4. Type 2 diabetic patients with ASCVD or high-risk cardiovascular risk factors (ASCVD includes acute coronary syndrome, stable coronary heart disease, revascularization, ischemic cardiomyopathy, ischemic stroke, transient ischemic attack, peripheral atherosclerotic disease. High-risk cardiovascular risk factors include age ≥55 years old, coronary artery/carotid artery/lower extremity artery stenosis >50%, or left ventricular hypertrophy)
5. Type 2 diabetic patients with CKD (eGFR30-60mL/min ·1.73m2)
6. Diabetic patients who are using SGLT2i to control blood glucose
7. Type 1 diabetes
8. Severe renal insufficiency (eGFR < 30mL/ min ·1.73m2), end-stage renal disease or dialysis patients
9. Previous diabetic ketoacidosis
10. Previous allergic reactions to SGLT2i
11. Severe hypoglycemia attacks in the past 12 months
12. Pregnant
13. Life expectancy less than 1 year
14. Subjects currently participating in other interventional clinical trials
15. Cardiac MRI contraindications (previous implantation of a metal device in the body) or refusal to undergo cardiac MRI
16. The researchers determine that there are factors that will affect the subjects' compliance with the intervention. Such as alcohol abuse, drug abuse, or behavioral disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in left atrial minimal volume index | 6 months
  Changes from baseline in left atrial minimal volume index in patients with AF treated with henagliflozin versus placebo using cardiac MRI.

SECONDARY OUTCOMES:
Atrial fibrillation quality of life | 6 months
  Changes from baseline in quality of life measured by the Atrial Fibrillation Effect on QualiTy of Life (AFEQT) survey. The AFEQT questionnaire has 20 items from 4 individual domains, including symptoms, daily activities, treatment concern, and treatment satisfaction. Each item is presented with a 7-point Likert response. Raw scores within each domain are transformed to a 0 to 100 scale, where a score of 0 indicates the most severe symptoms or disability and a score of 100 indicates no limitation or disability.
Change in left ventricular mass | 6 months
  Changes from baseline in LV mass as measured by cardiac MR in patients with AF treated with henagliflozin versus placebo.
Change in left ventricular end-diastolic volume index | 6 months
  Changes from baseline in LV end-diastolic volume index as measured by cardiac MR in patients with AF treated with henagliflozin versus placebo.
Change in left ventricular end-systolic volume index | 6 months
  Changes from baseline in LV end-systolic volume index as measured by cardiac MR in patients with AF treated with henagliflozin versus placebo.
Change in left ventricular global longitudinal strain | 6 months
  Changes from baseline in LV global longitudinal strain as measured by cardiac MR in patients with AF treated with henagliflozin versus placebo.
Change in left ventricular ejection fraction | 6 months
  Changes from baseline in LV ejection fraction as measured by cardiac MR in patients with AF treated with henagliflozin versus placebo.
Change in extracellular volume | 6 months
  Changes from baseline in extracellular volume (ECV) assessed using cardiac MR T1 mapping in patients with AF treated with henagliflozin versus placebo.
Change in left atrial ejection fraction | 6 months
  Changes from baseline in LA ejection fraction as measured by cardiac MR in patients with AF treated with henagliflozin versus placebo.
Change in left atrial global longitudinal strain | 6 months
  Changes from baseline in LA global longitudinal strain as measured by cardiac MR in patients with AF treated with henagliflozin versus placebo.
Change in right ventricular mass | 6 months
  Changes from baseline in RV mass as measured by cardiac MR in patients with AF treated with henagliflozin versus placebo.
Change in right atrial volume index | 6 months
  Changes from baseline in RA Volume Index as measured by cardiac MR in patients with AF treated with henagliflozin versus placebo.
Change in biomarkers of heart failure | 6 months
  Changes from baseline in biomarkers of heart failure (such as NT-proBNP) in patients with AF treated with henagliflozin versus placebo.
Change in 6min walk test | 6 months
  Changes from baseline in 6min walk test in patients with AF treated with henagliflozin versus placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Deyong Long, Principal Investigator — Beijing Anzhen Hospital; Changsheng Ma, Principal Investigator — Beijing Anzhen Hospital; Jianzeng Dong, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided